CLINICAL TRIAL: NCT01521663
Title: A Randomized, Double-Blind, Placebo-Controlled Safety and Efficacy Study of IPX159 in the Treatment of Moderate to Severe Restless Legs Syndrome (RLS)
Brief Title: Safety and Efficacy Study of IPX159 in Restless Legs Syndrome (RLS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPX159-B11-02
Record Dates: First submitted 2012-01-23; First posted 2012-01-31 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Restless Legs Syndrome
Keywords: Moderate to severe idiopathic RLS
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IPX159 (Experimental): IPX159 90 mg daily at week 1 with titration to 180 mg daily at week 2 with possible titration to 270 mg daily at week 3.
  Interventions: Drug: IPX159
- Sugar Pill (Placebo Comparator): IPX159 90 mg matching placebo daily at week 1 with titration to 180 mg matching placebo daily at week 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IPX159
  Arms: IPX159
Drug: Placebo
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to determine whether IPX159 is safe and effective in treating symptoms of RLS in subjects with Restless Legs Syndrome.

DETAILED DESCRIPTION:
IPX159 was developed as an extended release formulation to reduce the fluctuation in nefopam concentration compared to IR and to reduce the incidence of peak or rate related side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to sign an informed consent form (ICF) and Health Insurance Portability and Accountability Act (HIPAA) authorization
2. Males and females aged 18-70 with a history of primary RLS for ≥6 months prior to screening
3. Symptoms of RLS by medical history on at least 15 nights during the month prior to Screening
4. BMI 18.5-32
5. Negative alcohol and drug abuse screen
6. Negative serum pregnancy test
7. Agrees to use a medically acceptable method of contraception throughout the study and for 2 months after completing the study.
8. Able and willing to comply with the protocol, including availability for all scheduled clinic visits and telephone calls.

Exclusion Criteria:

1. Subjects who use or intend to use post screening the following medications or medication categories:

   * Sedative hypnotics, trazodone
   * Dopamine agonists, gabapentin, gabapentin enacarbil, pregabalin
   * Narcotic analgesics, other opioids, tramadol, cyclobenzaprine
   * Iron supplementation therapy
2. History of HIV, hepatitis B or C
3. Pregnant or breastfeeding.
4. History of or clinical signs of any form of epilepsy or seizures, excluding fever-related seizures in childhood.
5. History or presence of glaucoma
6. Planning to take herbal medications (eg, hypericum perforatum [St John's Wort], licorice, ephedra, ginkgo, ginseng) during the study.
7. Use of any investigational drug within the last 30 days or within a period of 5 times the drug's half-life, whichever is longer
8. Subjects who, in the opinion of the Investigator, should not participate in the study or are not capable of following the study schedule for any reason
9. Employees or family members of the Investigator, study site, the Sponsor, or Contract Research Organization (if any)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
International Restless Legs Syndrome Study Group (IRLSSG) Rating Scale | Assessed at each study visit (visits 1-7), an expected average of 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Principal Investigator — Impax Laboratories, Inc., acting through its Impax Pharmaceuticals Division (Impax)
Locations (38):
- United States (38):
  - University of Alabama at Birmingham, Brimingham, Alabama
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Scripps Clinic, La Jolla, California
  - Collaborative Neuroscience Network, Inc., Long Beach, California
  - The Research Center of Southern California, Oceanside, California
  - Stanford Center for Human Sleep Research, Redwood City, California
  - Neurological Research Institute, Santa Monica, California
  - Sleep-Alertness Disorder Center, Aurora, Colorado
  - PAB Clinical Research, Brandon, Florida
  - MD Clinical, Hallandale, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Resurgence Group, Palm Harbor, Florida
  - NeuroTrials Research Inc, Atlanta, Georgia
  - Georgia Health Sciences University, Augusta, Georgia
  - SleepMed of Central Georgia, Macon, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Community Research, Crestview Hills, Kentucky
  - Kentucky Research Group, Louisville, Kentucky
  - Johns Hopkins Bayview Medical Center Campus, Baltimore, Maryland
  - Sleep Health Centers, LLC, Brighton, Massachusetts
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - QUEST Research Institute, Farmington Hills, Michigan
  - Global Medical Institutes, LLC, Princeton, New Jersey
  - Fieve Clinical Research, Inc., New York, New York
  - Comprehensive Multiple Sclerosis Care Center, Patchogue, New York
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Community Research, Cincinnati, Ohio
  - Sleep Lab of Northeastern Pennsylvania, Clarks Summit, Pennsylvania
  - SleepMed of SC, Columbia, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - University of Tennesee Health Science Center, Memphis, Tennessee
  - Future Research Trials of Neurology, Austin, Texas
  - Clinical Trial Network, Houston, Texas
  - Bhupesh Dihenia, M.D., P.A., Lubbock, Texas
  - Paragon Research Center, LLC, San Antonio, Texas
  - Sleep Medicine Associates, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No